CLINICAL TRIAL: NCT01285427
Title: SeCore Sequencing Kit and 3500xl Dx Genetic Analyzer Clinical Performance Testing vs. SSP UniTray
Brief Title: Clinical Protocol SeCore, uTYPE and 3500 Dx System
Status: Completed | Type: Observational
Sponsor: Life Technologies Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DMR0000279
Record Dates: First submitted 2011-01-12; First posted 2011-01-28 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Human Leukocyte Antigens (HLA)
Keywords: DNA, sequencing; Identification and definition of Class I and II Human Leukocyte Antigens (HLA)

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — DNA isolated from whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DNA loci (SeCore vs. SSP UniTray platforms)

SUMMARY:
The purpose of this study is to compare the Invitrogen SeCore(R) sequencing system and uTYPE(R) interpretation software to the predicate device Invitrogen SSP UniTray(R) with UniMatch(R) interpretation software and show 95% concordance with 90% confidence.

DETAILED DESCRIPTION:
Testing will be performed on A, B, C, DRB1, DRB3/4/5, DQB1, and DPB1 loci. Additionally, testing will be performed using the following locus specific Group Specific Sequencing Primers: A, B, Cw, DPB1, DQB1 and DRB.

ELIGIBILITY:
Inclusion Criteria:

* Deidentified leftover blood samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A, B, C, DRB1, DRB3/4/5, DQB1, DPB1 loci
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Vella, Study Chair — Life Technologies

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not applicable. De-identified, archived whole blood samples
Period: Overall Study
Arm/Group | DNA Loci (SeCore vs. SSP UniTray Platforms)
Started | 300
Completed | 299 (One sample be discarded per FDA, sample drawn with heparin tube, not specified in protocol.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | DNA Loci (SeCore vs. SSP UniTray Platforms)
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Not Applicable, De-identified leftover blood samples
  Between 18 and 65 years | NA — Not Applicable, De-identified whole blood samples
  >=65 years | NA — Not Applicable, De-identified whole blood samples
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Not Applicable, de-identified leftover blood samples
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Not Applicable, De-identified leftover blood samples
  Male | NA — Not Applicable, De-identified leftover blood samples
de-identified whole blood samples [Number; unit: participants] | 300

OUTCOME MEASURES:

1. Primary Outcome: All SeCore® Kits,Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: All kits,the concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- Concordance: All SeCore Kits
Arm/Group | Concordance
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 99.6 [99.29 to 99.77]

2. Primary Outcome: SeCore® Kit, A Locus, Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: SeCore Kit, A Locus,the concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- Concordance: SeCore kit, A Locus
Arm/Group | Concordance
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 100.0 [99.01 to 100.0]

3. Primary Outcome: SeCore® Kit, B Locus (Single Amp), Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: SeCore® Kit, B Locus (Single Amp), The concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method.
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® Kit, B Locus (Single Amp): SeCore® Kit, B Locus (Single Amp)
Arm/Group | SeCore® Kit, B Locus (Single Amp)
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 99.7 [98.43 to 99.98]

4. Primary Outcome: SeCore® Kit, C Locus, Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: SeCore® Kit, C Locus, the concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method.
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® Kit, C Locus: SeCore® Kit, C Locus
Arm/Group | SeCore® Kit, C Locus
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 99.7 [98.43 to 99.98]

5. Primary Outcome: SeCore® Kit, DPB1 Locus, Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: SeCore® DPB1 Locus, the concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® DPB1 Locus Kit: SeCore® DPB1 Locus Kit
Arm/Group | SeCore® DPB1 Locus Kit
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 97.7 [95.65 to 98.90]

6. Primary Outcome: SeCore® Kit, DQB1 Locus, Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: the concordance rate was calculated and the corresponding exact two-sided 90% confidence interval was calculated by the Clopper-Pearson method
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® Kit, DQB1 Locus: SeCore® Kit, DQB1 Locus
Arm/Group | SeCore® Kit, DQB1 Locus
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 100.0 [99.01 to 100.0]

7. Primary Outcome: SeCore® Kit, DRB1 Locus, Primary Analysis of Concordance Rate (Clopper-Pearson CI)
Description: as for outcome 6
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® Kit, DRB1 Locus: SeCore® Kit, DRB1 Locus
Arm/Group | SeCore® Kit, DRB1 Locus
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 100.0 [99.01 to 100.0]

8. Primary Outcome: SeCore® Kit, DR Group Kit (DRB1 Locus), Primary Analysis of Concordance Rate (CI)
Description: as for outcome 6
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identifies leftover blood samples
Groups:
- SeCore® Kit, DR Group Kit (DRB1 Locus): SeCore® Kit, DR Group Kit (DRB1 Locus),
Arm/Group | SeCore® Kit, DR Group Kit (DRB1 Locus)
Number analyzed (Participants) | 299
Number analyzed (de-identifies leftover blood samples) | 299
percentage of concordant alleles | 100 [99.01 to 100.0]

9. Primary Outcome: SeCore® Kit, DR Group Kit (DRB345 Loci), Primary Analysis of Concordance Rate Clopper-Pearson CI)
Description: as for outcome 6
Time Frame: 10 weeks
Measure: Number (90% Confidence Interval); unit: percentage of concordant alleles
Units Other Than Participants: de-identified leftover blood samples
Groups:
- SeCore® Kit, DR Group Kit (DRB345 Loci): SeCore® Kit, DR Group Kit (DRB345 Loci),
Arm/Group | SeCore® Kit, DR Group Kit (DRB345 Loci)
Number analyzed (Participants) | 299
Number analyzed (de-identified leftover blood samples) | 299
percentage of concordant alleles | 99.7 [98.39 to 99.98]

ADVERSE EVENTS:
Arm/Group | Concordance
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No